CLINICAL TRIAL: NCT01555658
Title: Bivalirudin Plus Stenting in Long Lesion to Avoid Periprocedural Myocardial Necrosis Trial
Acronym: BILLION
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gennaro Sardella, Associate Professor in Cardiology, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BILLION
Record Dates: First submitted 2012-03-06; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Disease
Keywords: Long Lesions; Stent Implantation
MeSH Terms: conditions — Coronary Artery Disease | interventions — bivalirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bivalirudin (Experimental): Enrolled patients will be randomized 1:1 in the catheterization laboratory, after the decision to perform PCI by means of planned implantation of stents>33 mm in length in the same coronary vessel, to Bivalirudin
  Interventions: Drug: Bivalirudin
- Unfractioned Heparin (Experimental): Enrolled patients will be randomized in the catheterization laboratory, after the decision to perform PCI by means of planned implantation of stents>33 mm in length in the same coronary vessel, to Unfractioned Heparin.
  Interventions: Drug: Unfractioned Heparin

INTERVENTIONS:
Drug: Bivalirudin — Enrolled patients will be randomized 1:1 in the catheterization laboratory, after the decision to perform PCI by means of planned implantation of stents>33 mm in length in the same coronary vessel, to IV bivalirudin (0.75 mg/kg intravenous bolus followed by 1.75 mg/kg during procedure and 1.25mg/Kg infusion)
  Arms: Bivalirudin
Drug: Unfractioned Heparin — Enrolled patients will be randomized in the catheterization laboratory, after the decision to perform PCI by means of planned implantation of stents>33 mm in length in the same coronary vessel, to IV UFH (60 IU/kg intravenous bolus followed by boluses with target activated clotting time 200-250 s)
  Arms: Unfractioned Heparin

SUMMARY:
Background:

Randomized trials show improved outcomes among acute coronary syndrome (ACS) patients treated with Bivalirudin1. Optimal antithrombotic treatment in patients undergoing percutaneous coronary intervention (PCI) is crucial to balance the risk of post-PCI bleeding versus ischemic complications2. Bivalirudin, a direct thrombin inhibitor has been extensively investigated as an intra-procedural antithrombotic therapy in patients with stable angina, Non ST-segment elevation acute coronary syndrome (NSTE-ACS), and ST-segment elevation myocardial infarction (STEMI). Bivalirudin, when used with or without glycoprotein IIb/IIIa inhibitors (GPI) during PCI has been found to be superior to Unfractionated heparin (UFH) with or without GPI in reducing 30-day bleeding complications without significant increase in the rate of ischemic events3-5.

Moreover,after otherwise successful PCI,an increase in cardiac biomarkers has been shown to occur in 5% to 30% of patients6. Recent studies have focused their attention onthe reduction of infarct size and the incidence of periprocedural (type IVa) myocardial infarction (PMI)after elective PCI7-8. Therefore, we will perform a single-center, prospective and randomized study to assess if Bivalirudin versus UFHis effective in preventing elevation of biomarkers of MI after coronary stent implantation in patients already treated with aspirin and clopidogrel,with anatomically complex lesion.

Objective:

to assess the safety and efficacy of routine usage of the Bivalirudin vs UFH in patients with coronary artery disease (CAD), after stent implantation in coronary long lesions, to avoid periprocedural myocardial necrosis.

Setting:

Single-center, spontaneous, prospective, randomized 1:1 study of Bivalirudin infusion vs UFH in the setting of CAD, after PCI with stenting incoronary long lesions.

Comparison: Bivalirudin vs UFH, in preventing elevation of biomarkers of MI after coronary stent implantation in patients already treated with aspirin and clopidogrel, with anatomically complex lesion.

Population:Patients with diffuse CAD undergoing percutaneous treatment on a native coronary vessel with planned implantation stents in overlapping with a total stent length >33 mm for long coronary lesions in vessels with a reference vessel diameter 2.25-4.0 mm.

Assessment Following the procedure, blood samples for CK, CK-MB and Troponin will be collected at 6,12 and 24 h post PCI. CK-MB values will be considered abnormal if they will elevate above the upper limit of normal (ULN). This is set at 6 mg/L by our local laboratory. If the first blood sample showed a CK-MB level ≥18 mg/L (≥3 times upper normal limit), a second blood sample would be drawn every 8 h later until a downward trend will be observed. For patients with two or more blood samples drawn, the peak CK-MB level will be used for analysis.

End-points:

The primary end-point of this study will be the incidence of periprocedural myonecrosis that was defined as a peak post-procedural CK-MB elevation > 1 time the upper limit of normal (ULN) alone or associated with chest pain or ST-segment or T-wave abnormalities, in patients undergoing non-urgent PCI.

Secondary end-points will be the rate of MACCE (major adverse cerebro-cardiovascular events, ie the composite of death, myocardial infarction [defined according to the Academic Research Consortium statement], target vessel revascularization or stroke), the rate of major bleedings (Bleeding Academic Consortium [BARC] 3-5), minor bleedings (BARC 2), and the rate of NACE (net adverse clinical events, ie the composite of MACCE and major bleedings) at 30 days, 6 and 12 month follow-up. Adverse events will be determined by telephone interview and/or medical record review. Clinical follow-up: telephone-based interviews and office-based direct visits will be performed at 1, 6 and 12 months, respectively, for end-point adjudication.

Sample size and statistical analysis: Given an expected rate of abnormal post-procedural peak CK-MB > 1 x ULM of 48% (based on results of the INSTANT trial) for the control group and 29% for the experimental group (thus a 40% relative risk reduction), aiming for a 0.05 alpha and 0.80 power, a total of 204 patients will need to be enrolled (102 patients per group).

ELIGIBILITY:
Inclusion Criteria:Clinical Inclusion Criteria

Candidates for this study must meet all of the following criteria:

* Male or female able to understand and sign a witnessed informed consent
* Age ≥ 18 yo
* Patients with stable (CCS 1-4) or unstable angina pectoris (but with the most recent anginal episode occurring >48 hours before the index procedure) or documented silent ischemia
* Ongoing or recent episode (<48 hours) of unstable coronary artery disease (including non-ST-elevation acute coronary syndromes)
* Stable Hemodynamic conditions (systolic BP > 100 HR > 40 < 100).
* No clinical and ECG changes suggestive of ongoing acute or recent (<48 hours) myocardial infarction.

Angiographic inclusion criteria

* Angiographic evidence of a de novo lesion > 50% requiring implantation of two stents in overlapping with a total stent length> 33 mm and reference vessel diameter between 2.5 and 4.0 mm (by visual estimation) in one coronary vessel. Multiple lesions in the same vessels can be included but at least one lesion should require implantation of two stents in overlapping with a total stent length > 33 mm. The definition of multivessel disease requires an intention to treat at least two lesions (with a least one with the characteristics reported above) in two different major epicardial segments. For example, the presence of a lesion in the left anterior descending artery and in the obtuse marginal or the presence of a lesions in the right postero-lateral branch and in a diagonal branch will qualify as multivessel. The presence of lesions in the left anterior descending artery and in the diagonal branch will not qualify as multivessel. Bifurcation lesions and ostial lesions can be included, but only if at least two stent in overlapping with a total stent length > 33 mm are implanted in the same branch. When treating diffuse lesion in the same vessel, overlapping stenting is recommended with high pressure (>14 atm post-dilation) of the overlap zone. There is no maximum stent length to treat one coronary vessel.

Exclusion Criteria:

* Clinical Exclusion criteria

  * Female sex with childbearing potential
  * Age <18 years
  * Serum creatinine>2.5 mg/dl or with a creatinine clearance <40mL/min
  * Ongoing serious bleeding or bleeding diathesis
  * Previous stroke in the last 6 months
  * Major surgery within the previous 6 weeks
  * Platelet count <100,000 per mm3
  * Ejection Fraction below 30%
  * STEMIpatients' treated with primary-PCI, or rescue-PCI or facilitated-PCI or thrombolysis therapy.
  * Patients treated with Glycoprotein IIb/IIIa inhibitor for ACS
  * The patient has a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, or sensitivity to contrast which cannot be adequately pre-medicated.
  * Hemodynamic instability (systolic blood pressure < 100 mm Hg; heart rate < 40 bpm or >100 bpm; complex ventricular arrhythmias; AV block) requiring balloon counterpulsation or inotropic support.
  * The patient is simultaneously participating in another device or drug study. Patient must have completed the follow-up phase of any previous study at least 30 days prior to enrolment in this study.
  * Positive clinical history for intracranial neoplasia, AV malformation, aneurysm.
  * INR ≥ 2.0 or prothrombin time 1.2 times upper limit of normality
  * Clinically manifested reduced liver function
  * Programmed surgery within six months

Angiographic exclusion criteria

* Vessel size < 2.25 mm or > 5 mm (by visual estimation).
* Previous implantation of a bare-metal or drug-eluting stent in the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
The primary end point will be the rate of elevated post-procedural peak CK-MB mass ratio values above the upper limit of normal (ULN, defined as the ratio of the patient's peak value above the ULN) | 30 days
  The primary end-point of this study will be the incidence of periprocedural myonecrosis that was defined as a peak post-procedural CK-MB elevation > 1 time the upper limit of normal (ULN) alone or associated with chest pain or ST-segment or T-wave abnormalities, in patients undergoing non-urgent PCI.

SECONDARY OUTCOMES:
major adverse cerebro-cardiovascular events | 30 days - 6 and 12 months
  Secondary end-points will be the rate of MACCE (major adverse cerebro-cardiovascular events, ie the composite of death, myocardial infarction [defined according to the Academic Research Consortium statement]
major and minor bleedings | 30 days, 6 and 12 months
  In according with Bleeding Academic Consortium (BARC classification)
the rate of net adverse clinical events (NACE) | 30 days, 6 and 12 months
  the composite of MACCE and major bleedings

CONTACTS AND LOCATIONS:
Locations (1):
- Dept.of Cardiovascular Sciences Policlinico Umberto I, Rome, Italy